CLINICAL TRIAL: NCT03426072
Title: Safer Care for Older People in (Residential) Environments
Acronym: SCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: SCOPE ABBC
Record Dates: First submitted 2018-02-01; First posted 2018-02-08 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2021-04

CONDITIONS: Nursing Homes
Keywords: quality improvement

STUDY DESIGN:
Intervention Model Description: cluster randomised controlled trail with nursing home unit as the cluster, care aides and residents as the unit of analysis
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: control sites are propensity matched to intervention sites. All sites have comprehensive dataset. Trial status of each home is unknown to assessor and statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified IHI breakthrough series (Experimental): The SCOPE intervention is a complex, "high facilitation", multi-component intervention operating at the microsystem (resident care unit) level of the organization and is designed to engage, develop, and equip Health Care Aides to implement improvement initiatives.
  Interventions: Other: modified IHI breakthrough series
- Control (No Intervention): The control units (propensity matched) have no intervention and form a naturalistic control

INTERVENTIONS:
Other: modified IHI breakthrough series — There are five main elements to the intervention:
  1. Establishment of the team and set up
  2. Establishing baseline performance and knowledge
  3. Ongoing developmental support
  4. Learning sessions (3)
  5. Action periods (3)
  6. The actual facilitative actions (e.g., coaching, guiding, mentoring, supporting) occur in combination with limited teaching, largely during telephone conferences but also in any visit, which may occur up to quarterly.
  5. The concluding session is an opportunity for networking, sharing successes and making plans for the continuation of project work following the end of formal support
  Arms: modified IHI breakthrough series

SUMMARY:
The overall aim of the program is to advance knowledge translation science in order to improve clinical and staff related outcomes in long term care facilities (nursing homes) in western Canada. SCOPE will assess the effect of Care Aide led Quality Improvement efforts on staff quality of work life as well as resident quality of care. A key element of SCOPE is a leadership development stream which introduces complexity science and education on quality improvement which aims to support front line teams with their improvement initiative

DETAILED DESCRIPTION:
The aim of this study is to assess the effects of a facilitation-based improvement intervention on three primary performance outcomes: (1) staff reported use of best practices, (2) measures of staff work engagement and job satisfaction, and (3) resident quality of care. Within the context of the Translating Research in Elder Care study (Pro00037937), the influence of staff characteristics related to work performance and unit context scores (leadership, culture, resources) on the three primary outcomes will be assessed Background Translating Research in Elder Care (TREC) is an ongoing applied research program that began in 2007. TREC is focused on practical solutions that will improve quality of care provided to nursing home residents, enrich the work life of their caregivers, and enhance system efficiencies and effectiveness. In TREC 1, teams of researchers worked together with decision makers from the residential long term care (LTC) sector on multiple studies in Manitoba, Saskatchewan, Alberta and to a lesser extent, British Columbia (SCOPE pilot only). Data were collected from approximately 4000 care providers and residents using the Resident Assessment Index Minimum data Set (RAI-MDS) 2.0 in participating TREC nursing homes.

TREC has already established its value to the health system by demonstrating improvements in resident care, clinical outcomes, and staff well-being. Information data collected from over 100,500 resident assessments combined with the staff and facility surveys now forms the TREC Measurement System (TMS Project). This wealth of data has informed the SCOPE pilot project in 2010 and SCOPE was conceived as a result of this data.

The SCOPE intervention is designed as a randomized controlled trial (RCT). For our primary outcome measure (change in Conceptual Research Use (CRU)between pre and post intervention periods) a sample size of 34 units per arm is adequate to detect an effect size of 0.67 or greater (using the standard deviation for the change in CRU between pre and post intervention periods for intervention and non-intervention from the SCOPE pilot data at 80% power, with an alpha 0.05, for a 2-tailed comparison of independent samples. The intervention will take place in as many as 45 of the facilities involved in the TMS project (Pro00037937) to take account of drop -outs. Each facility will have a Senior Sponsor (generally the Director of Care or Exec Director). Participants in the intervention teams will be from a single unit in each intervention facility and will include 3 Health Care Aides who will lead the team, as well as 2 other members of that unit which can include other allied professional staff, nurses, and Occupational Therapist /Rec Aides. One member of the team must be the Team sponsor (generally the unit's care manager) removes obstacles for the team.

ELIGIBILITY:
Inclusion Criteria:

Facilities must be a part of TMS to be eligible for SCOPE. This means that they are:

* A nursing home or residential long term care facility which provides 24-hour on-site housing and health care services care for older adults by professional (nursing) staff and others
* Registered with the provincial government
* 90% of residents aged 65 or over
* RAI-MDS 2.0 implemented since January 2011
* Facility operations conducted in the English language
* Urban* facilities located within designated health regions and within 110 km of the TREC-designated hub for the health region:

  * Fraser Health Authority (Hub is New Westminster)
  * Interior Health Authority (Hubs are Kelowna, Kamloops)
  * Alberta (AHS): Edmonton and Calgary Zones (Edmonton & Calgary are hubs)

Exclusion Criteria:

* Facilities that have participated in the SCOPE pilot study (Pro00012517)
* Facilities integrated with acute care. Defined as residential long-term care facility (usually one or more resident units) that:

  * Are physically located within an acute care facility and
  * Share central services (e.g., human resources, laundry), as well as, other functions integral to care delivery such as staffing, supervision, performance management, etc.)
  * Co-located services (where the daily operations of the resident units are managed separately and staff independently) are acceptable
* Facilities with more than one sub-acute (e.g., orthopaedic rehab) unit
* Facilities with fewer than 35 long-term care beds
* Facilities which are expected to undergo major change within the next two years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Conceptual Research Use | 1 year
  Conceptual use of best practices: indirect measure of application of research and best practices measured by a 5 item scale. BMC Health Services Research 2011; 11:107 demonstrating acceptable validity and reliability

SECONDARY OUTCOMES:
Resident Assessment Index -minimal Data Set (RAI-MDS) factors | change between intervention and control groups 1 year post intervention
  Resident outcome data obtained from quarterly RAI-MDS 2.0 reports, examined as the change in the quality indicator worked upon (e.g., pressure ulcers, pain, declining behaviour) between baseline and study end
Staff outcomes | change between intervention and control groups 1 year post intervention
  Staff (healthcare aide) outcomes of work engagement, burnout, empowerment, organizational citizenship behaviours and job satisfaction. We will assess baseline performance using the Rantz Observable Indicators of Quality survey

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
the data will be made available on request according to TREC data sharing policies

REFERENCES:
- [Derived] Wagg A, Hoben M, Ginsburg L, Doupe M, Berta W, Song Y, Norton P, Knopp-Sihota J, Estabrooks C. Safer Care for Older Persons in (residential) Environments (SCOPE): a pragmatic controlled trial of a care aide-led quality improvement intervention. Implement Sci. 2023 Mar 29;18(1):9. doi: 10.1186/s13012-022-01259-8. PMID 36991434